CLINICAL TRIAL: NCT00020891
Title: The Use Of Multiple CT Scans To Reduce Target Positioning Errors In Patients Undergoing External Beam Radiotherapy Treatment For Prostate Cancer
Brief Title: CT Scans in Guiding the Treatment of Patients With Prostate Cancer Who Are Undergoing Radiation Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Diagnostic
Other Study IDs: 01-022; P30CA008748 (NIH); MSKCC-01022; NCI-G01-1968
Record Dates: First submitted 2001-07-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

INTERVENTIONS:
Procedure: computed tomography
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Multiple CT scans may improve the accuracy of radiation therapy for prostate cancer.

PURPOSE: Phase I trial to study the effectiveness of multiple CT scans in guiding the treatment of patients who have prostate cancer and are undergoing radiation therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the accuracy of radiotherapy delivery using multiple CT scans to guide patient positioning vs the standard portal image guided procedure in patients with prostate cancer undergoing external beam radiotherapy.
* Determine the reduction in the proportion of patients with large target positioning errors using the CT-guided procedure.
* Determine organ motion and setup errors over the course of radiotherapy in order to develop efficient clinical intervention strategies in these patients.

OUTLINE: Patients undergo radiotherapy over 9 weeks. Patients undergo a CT scan immediately prior to receiving radiotherapy on treatment days 3-8 and then weekly thereafter. On 3 different days, patients also undergo CT scan immediately after radiotherapy. If the CT scans indicate a correction that exceeds the action level currently in effect, then beginning with the next treatment, the patient's position with respect to the radiation field is adjusted.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Undergoing external beam intensity-modulated radiotherapy for prostate cancer
* Able to maintain treatment position for about 40 minutes

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics

Surgery:

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2001-03; Primary Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Treatment accuracy

SECONDARY OUTCOMES:
Reduction in the proportion of patients with large target positioning errors using CT guided procedure
Organ motion and setup errors

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lovelock, PhD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States